CLINICAL TRIAL: NCT02104882
Title: INTRAGO-Intraoperative Radiotherapy for Glioblastoma - a Phase I/II Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Frederik Wenz, Director, Department of Radiation Oncology, Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTRAGO-I/II
Record Dates: First submitted 2014-03-26; First posted 2014-04-07 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; High-Grade Glioma; Malignant Glioma; IORT
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraoperative Radiotherapy (Experimental): Following conventional frameless neuronavigation-guided microsurgical tumor resection, patients will receive IORT with 20-40 Gy (prescribed to the applicator surface). Not later than 4 weeks, radiochemotherapy (RCT) will be initiated, consisting of a total EBRT dose of 60 Gy (delivered in fractions of 2 Gy) and concomitant chemotherapy with temozolomide (50 mg/m2/d). Four weeks after RCT, cycling chemotherapy with temozolomide (150-200mg/m2/d/cycle) will be applied.
  Interventions: Radiation: Intraoperative Radiotherapy (Applicator Surface Dose: 20-40 Gy)

INTERVENTIONS:
Radiation: Intraoperative Radiotherapy (Applicator Surface Dose: 20-40 Gy)

SUMMARY:
Glioblastoma multiforme (GBM) is a disease with an extremely poor prognosis. Despite surgery and radiochemotherapy, the tumors are likely to grow back very quickly.

Intraoperative radiotherapy (IORT) may improve local control rates while sparing healthy tissue (Giordano et al. 2014). IORT takes place before cranioplasty directly after gross (or subtotal) tumor resection. Several past studies on IORT for GBM conducted in Japan and Spain have yielded encouraging results (Sakai et al. 1989; Matsutani et al. 1994; Fujiwara et al. 1995; Ortiz de Urbina et al. 1995).

However, the full potential of the procedure is to date largely unexplored as most previous studies used forward-scattering (electron-based) irradiation techniques, which frequently led to inadequately covered target volumes. With the advent of the spherically irradiation devices such as the Intrabeam® system (Carl Zeiss Meditec AG, Oberkochen, Germany), even complex cavities can be adequately covered with irradiation during IORT. However, there is no data on the maximum tolerated dose of IORT with low-energy X-rays as generated by this system.

The INTRAGO I/II study aims to find out which dose of a single shot of radiation, delivered intraoperatively direct after surgery, is tolerable for patients with GBM. A secondary goal of the study is to find out whether the procedure may improve survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme in frozen sections
* Age ≥50 years
* Karnofsky Performance Index ≥ 50%
* Informed consent
* Adequate birth control (e.g., oral contraceptives)

Exclusion Criteria:

* Astrocytoma ≤ WHO grade III
* Gliomatosis cerebri
* Multifocal lesions
* Infratentorial localization
* Previous cranial radiation therapy (any location)
* Uncontrolled intercurrent illnesses including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Contraindications for general anaesthesia
* Bleeding or clotting disorders
* Contraindications for MRI or CT scans
* Pregnant or breastfeeding women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 3 Months
  The maximum tolerated (single) dose of IORT with 50 kV X-rays will be assessed using a classical "3+3" design:
  The first cohort of 3 patients will receive IORT with 20 Gy (prescribed to the applicator surface). If none of these patients experiences a DLT, another three patients will be treated at the next higher dose level (30 Gy). However, should a patient experience a DLT, 3 more patients will be treated at the same dose level. The dose escalation stops if two ore more patients in a cohort of 3-6 patients experience DLT. The MTD is then defined as the dose level just below the toxic dose level.
  Two types of DLT are defined:
  Early DLT (≤ 3 weeks after IORT):
  * wound infections / wound healing difficulties requiring surgical intervention
  * IORT-related cerebral bleeding or ischemia
  Delayed DLT (≤ 3 months after IORT):
  * Symptomatic brain necrosis requiring surgical intervention
  * Early termination of EBRT (before the envisaged dose of 60 Gy) due to radiotoxicity

SECONDARY OUTCOMES:
Progression Free Survival | 3 Years
Overall Survival | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Wenz, MD, Study Chair — Department of Radiation Oncology, Universitätsmedizin Mannheim, University of Heidelberg; Peter Schmiedek, MD, Principal Investigator — Department of Neurosurgery, Universitätsmedizin Mannheim, University of Heidelberg
Locations (1):
- Universitätsmedizin Mannheim, University of Heidelberg, Mannheim, Germany

REFERENCES:
- [Background] Giordano FA, Brehmer S, Abo-Madyan Y, Welzel G, Sperk E, Keller A, Schneider F, Clausen S, Herskind C, Schmiedek P, Wenz F. INTRAGO: intraoperative radiotherapy in glioblastoma multiforme-a phase I/II dose escalation study. BMC Cancer. 2014 Dec 22;14:992. doi: 10.1186/1471-2407-14-992. PMID 25535398
- [Background] Matsutani M, Nakamura O, Nagashima T, Asai A, Fujimaki T, Tanaka H, Nakamura M, Ueki K, Tanaka Y, Matsuda T. Intra-operative radiation therapy for malignant brain tumors: rationale, method, and treatment results of cerebral glioblastomas. Acta Neurochir (Wien). 1994;131(1-2):80-90. doi: 10.1007/BF01401457. PMID 7709789
- [Background] Sakai N, Yamada H, Andoh T, Takada M, Hirata T, Funakoshi T, Doi H, Yanagawa S. [Intraoperative radiation therapy for malignant glioma]. Neurol Med Chir (Tokyo). 1989 Apr;29(4):312-8. doi: 10.2176/nmc.29.312. Japanese. PMID 2478913
- [Background] Fujiwara T, Honma Y, Ogawa T, Irie K, Kuyama H, Nagao S, Takashima H, Hosokawa A, Ohkawa M, Tanabe M. Intraoperative radiotherapy for gliomas. J Neurooncol. 1995;23(1):81-6. doi: 10.1007/BF01058463. PMID 7623073
- [Background] Ortiz de Urbina D, Santos M, Garcia-Berrocal I, Bustos JC, Samblas J, Gutierrez-Diaz JA, Delgado JM, Donckaster G, Calvo FA. Intraoperative radiation therapy in malignant glioma: early clinical results. Neurol Res. 1995 Aug;17(4):289-94. doi: 10.1080/01616412.1995.11740329. PMID 7477745